CLINICAL TRIAL: NCT03455322
Title: Pros & Cons of Norepinephrine Infusion Versus Midodrine & Octreotide in Patients With Hepatorenal Syndrome Type 1 in Intensive Care Unit.
Brief Title: Norepinephrine Infusion Versus Midodrine & Octreotide in Patients With Hepatorenal Syndrome Type 1.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, Consultant of Intensive care medicine, Ph D, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHTMRI-2
Record Dates: First submitted 2018-01-03; First posted 2018-03-06 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Renal Impairment in Hepatorenal Syndrome
MeSH Terms: interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- norepinephrine (Active Comparator): norepinephrine continuous intravenous infusion in a dose of 0.05-0.3ug/Kg/min. average7-10 days to keep mean arterial pressure ≥ 80-100mmHg & continued either until HRS reversal or for maximum 10 days.
  Interventions: Drug: norepinephrine versus midodrine & octreotide
- midodrine & octreotide (Active Comparator): midodrine 5mg three times/day orally & can be increased every 24h up to 12.5mg three times daily plus octreotide 100ug/ 6h subcutaneous & if needed increased to 200ug/6hS.C. for 7-10 days
  Interventions: Drug: norepinephrine versus midodrine & octreotide

INTERVENTIONS:
Drug: norepinephrine versus midodrine & octreotide — either intravenous infusion (IVi) norepinephrine in a dose of 0.05-0.3ug/Kg/min. to keep mean arterial pressure ≥ 80-100mmHg & continued either until HRS reversal or for maximum 10 days or oral midodrine 5mg three times/day & can be increased every 24h up to 12.5mg three times daily plus octreotide 100ug/ 6h subcutaneous & if needed increased to 200ug/6h.

SUMMARY:
This study aimed to investigate the efficacy of midodrine plus octreotide versus norepinephrine and to determine the predictive factors of response in patients with HRS-AKI.

DETAILED DESCRIPTION:
Both sexes aged 18 years or older having cirrhosis, ascites, and a diagnosis of HRS-AKI based on the 2015 International Club of Ascites (ICA) diagnostic criteria [2] were eligible for participation.

Screening and eligibility criteria were verified upon admission to the ICU. A diagnosis of AKI was established through comparing sCr value at time of ICU admission to that recorded in the patient's file. Patients who meet all other diagnostic criteria of HRS-AKI provided by the previous definition [2] were enrolled in the study. Qualified patients were subjected to baseline assessments after informed consent signature. It included vital sign measurements, presence of comorbidities, height and weight, Child-Pugh score and Sequential Organ Failure Assessment (SOFA) score. Vital signs, Blood urea nitrogen, sCr, serum sodium, serum albumin, total bilirubin, and complete blood count with differential were measured at baseline and at daily basis throughout the study period. Patients were randomized in a 1:1 ratio to receive either continuous infusion of norepinephrine in an initial dose of 0.5mg/h (Maximum 3 mg/h or oral midodrine 5mg three times/day (Maximum 12.5mg three times/day) plus octreotide 100μg/6h as subcutaneous injection (Maximum 200 μg/6h). Duration of treatment was allowed to extend to a maximum of 10 days. Administration of albumin at doses of 20 to 40 gm/day was recommended, as clinically indicated, for all patients in both study arms as per current ICA guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All patients that will be included in the study have cirrhosis as diagnosed by clinical, biochemical, and ultrasound findings, with HRS type 1, the absence of bacterial infections; however, patients with bacterial infections could be included in the study if renal failure persisted after infection resolution by clinical, laboratory indices up to 48 hours.

Exclusion Criteria:

* Patients will be excluded if there are advanced cardiovascular diseases due to poor prognosis or any extrahepatic disease that could affect the short-term prognosis, the presence of advanced hepatocellular carcinoma or presence of contraindication to norepinephrine as hypotension due to blood volume deficits except emergency measure, mesenteric or peripheral vascular thrombosis unless there is life-saving procedure, profound hypoxia or hypercarbia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
the proportion of patients achieved full response | within10 days
  defined as return of sCr to a value within 0.3 mg/dl of the baseline value

SECONDARY OUTCOMES:
the proportion of patients achieved partial response | within 10 days
  defined as a regression of at least one AKI stage with a fall in the sCr value to ≥0.3 mg/dl above the baseline value
Incidence of HRS reversal | within 10 days
  defined as at least one sCr value of ≤ 1.5 mg/dl while on treatment
incidence of HRS-AKI relapse | 30 days
  relapse of HRS-AKI after cessation of treatment
overall survival | 30 days
  patients who are survived
adverse events experienced throughout the study period in both treatment groups. | within 10 days
  The incidence of hepatic encephalopathy episodes, bacterial infections, gastrointestinal bleeding, myocardial infarction, arrhythmia, circulatory overload and arterial hypertension was assessed at the end of the study. The need for mechanical ventilation and the need for dialysis.

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 - 12 months

REFERENCES:
- [Derived] El-Desoki Mahmoud EI, Abdelaziz DH, Abd-Elsalam S, Mansour NO. Norepinephrine is More Effective Than Midodrine/Octreotide in Patients With Hepatorenal Syndrome-Acute Kidney Injury: A Randomized Controlled Trial. Front Pharmacol. 2021 Jul 2;12:675948. doi: 10.3389/fphar.2021.675948. eCollection 2021. PMID 34276366